CLINICAL TRIAL: NCT04171921
Title: Robotic Versus Open Primary Ventral Hernia Repair: a Randomized Controlled Trial
Brief Title: Robotic Versus Open Primary Ventral Hernia Repair
Acronym: Robovent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Dr Jonathan Douissard, Staff surgeon visceral surgery department, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-00113
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Ventral Hernia
Keywords: Open ventral hernia repair; Robotic ventral hernia repair; Surgical site complications; Esthetic satisfaction; Pain; Pain-killers consumption; Costs; Operative time; Early hernia recurrence; General complications
MeSH Terms: conditions — Hernia, Ventral; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic ventral hernia repair (Active Comparator)
  Interventions: Procedure: Robotic ventral hernia repair
- Open ventral hernia repair (Active Comparator)
  Interventions: Procedure: Open ventral hernia repair

INTERVENTIONS:
Procedure: Robotic ventral hernia repair — Laparoscopic robotically assisted trans-abdominal pre-peritoneal epigastric or umbilical hernia repair with closure of fascial defect and non-adsorbable mesh reinforcement
  Arms: Robotic ventral hernia repair
Procedure: Open ventral hernia repair — Standard open pre-peritoneal epigastric or umbilical hernia repair with closure of fascial defect and non-adsorbable mesh reinforcement
  Arms: Open ventral hernia repair

SUMMARY:
Umbilical and epigastric hernia repair, whether considering primary or incisional hernias, are associated with a high risk of local complications, with global rate of surgical complications at one month up to 25%. To date three techniques are used.

Open ventral hernia repair (OVHR) is associated with a high risk of surgical site infection, wound dehiscence, and hematoma, but is the main technique due to advantages such as cost-effectiveness, short operative time and totally extra-peritoneal repair.

Laparoscopic hernia repair (LHR) reduces these complications but implies to place a mesh in intra-peritoneal position which is known to lead to adhesions, requires advanced laparoscopic skills, does not allow the closure of the defect due to limited range of motion, and can lead to excessive pain and pain-killers consumption due to the use of "tackers" to hold the mesh in place.

Robotic ventral hernia repair (RVHR) uses the same laparoscopic access as LHR but thanks to the extended range of motion given by the robotic system allows defect closure, pre-peritoneal placement of the mesh and requires less technical skills.

LHR is of very low adoption in Geneva University Hospital for the aforementioned inconvenient. Moreover, the final result of the procedure is not the same than with OVHR or RVHR, since the defect is not primarily closed and the mesh is in intra-peritoneal position. OVHR and RVHR , however, lead to the same final result and only defer by the access type (direct vs. laparoscopic). RVHR is gaining rapid popularity and adoption in the United States but remains a costly solution. It is unclear whether the supposed benefits for the patients of RVHR overwhelm the extra costs and time, especially by reducing the complication rate and consecutive in-hospital and out-hospital costs. Moreover, increasing experience of the robotic system in Geneva University Hospital has led to a significant costs and time reduction in other robotic procedures and could eventually make RVHR cost effective if its clinical benefits were to be proven.

This study aims at demonstrating that robotic trans-abdominal pre-peritoneal (rTAPP) primary ventral hernia repair leads to lower surgical site complication rate than the same procedure performed through standard open approach (OVHR), while being an acceptable solution from an economic, operative time and functional standpoint.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent as documented by signature
* Aged 18 years or older
* Undergoing primary umbilical or epigastric hernia repair of size between 1cm and 5cm +/-5mm, with mesh reinforcement, in the Visceral Surgery Department of the University Geneva Hospital

Exclusion Criteria:

* Patients under corticosteroids or other immunosuppressive treatment
* Pregnancy or breastfeeding
* Intention to become pregnant during the course of the study
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential
* Incisional hernia and/or substantial history of intra-abdominal surgery
* Upon anesthesiologist evaluation, clinically significant concomitant disease states which require to shorten operative time at maximum
* Upon anesthesiologist evaluation, clinically significant concomitant disease states being a contra-indication to laparoscopic approach and/or general anesthesia
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Surgical site complication | At 31 days after surgery
  Yes or no

SECONDARY OUTCOMES:
Detailed surgical site complications | At 31 days after surgery
  Classified according to aforementioned Clavien-Dindo's scoring system (scale from 1 to 5, higher score mean a worse outcome)
General complications, not directly related to surgical site | At 31 days after surgery
  Classified according to aforementioned Clavien-Dindo's scoring system (scale from 1 to 5, higher score mean a worse outcome)
General pain: Visual Analogue Scale | At 31 days after surgery
  Evaluated using Visual Analogue Scale (VAS, scale from 0 to 10, higher score mean a worse outcome))
Painkillers consumption | At 31 days after surgery
  Recorded from patient's medical record for in-hospital stay for out-hospital period will be evaluated with consumption recall at each visit
Esthetic satisfaction: European Hernia Society Quality of Life (EuraHS-QoL) | At 31 days after surgery
  Using European Hernia Society Quality of Life (EuraHS-QoL) ( scale from 0-90, with the lower scores being the most favorable outcome)
Quality of life score | At 31 days after surgery
  Using European Hernia Society Quality of Life (EuraHS-QoL) form (scale from 0-90, with the lower scores being the most favorable outcome)
In-hospital costs | At day 31 after surgery
  Hospitalization costs including medications, care and labs, cost of the procedure, diagnosis related group class, total amount billed to the insurance.
  Derived using REKOLE® method.
Out-hospital costs | At day 31 after surgery
  Consults and drugs Estimated based on hospital's billing data.
Early recurrence at 1 month | At day 31 after surgery
  Evaluated by physical evaluation
Defect size | During surgery
  Measured with ruler
Number of device related adverse events by the operating surgeon | During surgery
  Surgical complications which are identified by the operating surgeon as directly related to malfunction of the robotic system

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Douissard, MD, Principal Investigator — University of Geneva, Geneva University Hospital
Locations (1):
- Visceral surgery department - Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poulose BK, Shelton J, Phillips S, Moore D, Nealon W, Penson D, Beck W, Holzman MD. Epidemiology and cost of ventral hernia repair: making the case for hernia research. Hernia. 2012 Apr;16(2):179-83. doi: 10.1007/s10029-011-0879-9. Epub 2011 Sep 9. PMID 21904861
- [Background] Holihan JL, Alawadi Z, Martindale RG, Roth JS, Wray CJ, Ko TC, Kao LS, Liang MK. Adverse Events after Ventral Hernia Repair: The Vicious Cycle of Complications. J Am Coll Surg. 2015 Aug;221(2):478-85. doi: 10.1016/j.jamcollsurg.2015.04.026. Epub 2015 May 9. PMID 26206646
- [Background] Bisgaard T, Kehlet H, Bay-Nielsen M, Iversen MG, Rosenberg J, Jorgensen LN. A nationwide study on readmission, morbidity, and mortality after umbilical and epigastric hernia repair. Hernia. 2011 Oct;15(5):541-6. doi: 10.1007/s10029-011-0823-z. Epub 2011 May 3. PMID 21538150
- [Background] Helgstrand F. National results after ventral hernia repair. Dan Med J. 2016 Jul;63(7):B5258. PMID 27399983
- [Background] Reynolds D, Davenport DL, Korosec RL, Roth JS. Financial implications of ventral hernia repair: a hospital cost analysis. J Gastrointest Surg. 2013 Jan;17(1):159-66; discussion p.166-7. doi: 10.1007/s11605-012-1999-y. Epub 2012 Sep 11. PMID 22965649
- [Background] Hajibandeh S, Hajibandeh S, Sreh A, Khan A, Subar D, Jones L. Laparoscopic versus open umbilical or paraumbilical hernia repair: a systematic review and meta-analysis. Hernia. 2017 Dec;21(6):905-916. doi: 10.1007/s10029-017-1683-y. Epub 2017 Oct 14. PMID 29032495
- [Background] Froylich D, Segal M, Weinstein A, Hatib K, Shiloni E, Hazzan D. Laparoscopic versus open ventral hernia repair in obese patients: a long-term follow-up. Surg Endosc. 2016 Feb;30(2):670-675. doi: 10.1007/s00464-015-4258-y. Epub 2015 Jun 20. PMID 26091995
- [Background] Muysoms FE, Bontinck J, Pletinckx P. Complications of mesh devices for intraperitoneal umbilical hernia repair: a word of caution. Hernia. 2011 Aug;15(4):463-8. doi: 10.1007/s10029-010-0692-x. Epub 2010 Jun 17. PMID 20556448
- [Background] Liang MK, Berger RL, Li LT, Davila JA, Hicks SC, Kao LS. Outcomes of laparoscopic vs open repair of primary ventral hernias. JAMA Surg. 2013 Nov;148(11):1043-8. doi: 10.1001/jamasurg.2013.3587. PMID 24005537
- [Background] Tandon A, Pathak S, Lyons NJ, Nunes QM, Daniels IR, Smart NJ. Meta-analysis of closure of the fascial defect during laparoscopic incisional and ventral hernia repair. Br J Surg. 2016 Nov;103(12):1598-1607. doi: 10.1002/bjs.10268. Epub 2016 Aug 22. PMID 27546188
- [Background] Hilling DE, Koppert LB, Keijzer R, Stassen LP, Oei IH. Laparoscopic correction of umbilical hernias using a transabdominal preperitoneal approach: results of a pilot study. Surg Endosc. 2009 Aug;23(8):1740-4. doi: 10.1007/s00464-008-0177-5. Epub 2008 Nov 18. PMID 19015918
- [Result] Colavita PD, Tsirline VB, Belyansky I, Walters AL, Lincourt AE, Sing RF, Heniford BT. Prospective, long-term comparison of quality of life in laparoscopic versus open ventral hernia repair. Ann Surg. 2012 Nov;256(5):714-22; discussion 722-3. doi: 10.1097/SLA.0b013e3182734130. PMID 23095614
- [Derived] Douissard J, Meyer J, Dupuis A, Peloso A, Mareschal J, Toso C, Hagen M. Robotic versus open primary ventral hernia repair: A randomized controlled trial (Robovent Trial). Int J Surg Protoc. 2020 Apr 4;21:27-31. doi: 10.1016/j.isjp.2020.03.004. eCollection 2020. PMID 32368702